CLINICAL TRIAL: NCT00001645
Title: Evaluation, Treatment, and Monitoring of Patients With Known or Suspected Parasitic Infection
Brief Title: Evaluation, Treatment and Monitoring of Patients With a Known or Suspected Parasitic Infection
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970096; 97-I-0096
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01-16

CONDITIONS: Malaria; Intestinal Worms; GI Protozoa; Echiniococcus; Strongyloides
Keywords: Helminth Infection; Parasite; Known Parasitic Infection; Suspected Parasitic Infection; Natural History
MeSH Terms: conditions — Malaria; Trematode Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Diarrhea GI parasite: Subjects infected with a GI parasite
- Echinococcus: Subjects infected with echinococcus
- Intestinal worm: Subjects infected with parasitic intestinal worm
- Malaria: Subjects infected with malaria
- Parasitic infection: Subjects infected with a parasitic infection that is not included in the other cohorts

SUMMARY:
The purpose of this study is to evaluate, treat and follow patients with parasitic infections.

People with a known or suspected parasitic infection who are at least 1 year old may be enrolled. This study does not involve any experimental treatments.

Participants will have a physical examination and laboratory tests on blood, stool, or urine. Blood samples may be collected at regular intervals, but no more than 450 ml (15 ounces) of blood will be drawn from adults, and no more than 7 ml (1-1/2 teaspoons) per kg (2.2 pounds) of body weight from children, in any 6-week period. Other tests may include x-rays, electrocardiogram (EKG), or tissue biopsy (surgical removal of a small tissue sample), depending on the individual s condition.

Patients may be offered treatment or may be referred to another study that is more appropriate for the problem. Any treatment provided in this study will be according to standard medical practice for the patient s specific medical problem. Patients responses to treatment will be evaluated at regularly scheduled clinic visits. The length of time between visits and the total duration of the study for a given individual will be determined by the study doctor, based on that person s medical condition.

DETAILED DESCRIPTION:
This study is designed as a prospective study to evaluate and treat patients with parasitic infection. Patients with known or suspected parasitic infection will be enrolled and will be evaluated for the presence of a parasitic infection. Minimal studies scheduled for each visit will include a medical history, physical examination, routine laboratory tests, and specialized diagnostic procedures for possible parasitic infections. Treatment plans will be individualized for each patient's particular condition, and the number and length of additional visits and diagnostic evaluations will vary accordingly. Specific treatment regimens will be in accordance with standard medical practice.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 3 or over.

Access to a primary medical care provider outside of the NIH

Clinical evidence suggestive of a parasitic infection

EXCLUSION CRITERIA:

Less than 3 years of age

No evidence suggestive of a parasitic infection

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 1998-10-10 (Actual)

PRIMARY OUTCOMES:
The Laboratory of Parasitic Diseases has been conducting studies of the diagnosis, treatment, and pathogenesis of wide variety of parasitic infections. | 1 year
  Elimination of parasitic infection.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Nutman TB. Human infection with Strongyloides stercoralis and other related Strongyloides species. Parasitology. 2017 Mar;144(3):263-273. doi: 10.1017/S0031182016000834. Epub 2016 May 16. PMID 27181117
- [Background] O'Connell EM, Nutman TB. Eosinophilia in Infectious Diseases. Immunol Allergy Clin North Am. 2015 Aug;35(3):493-522. doi: 10.1016/j.iac.2015.05.003. PMID 26209897
- [Background] Nash TE, Ohl CA, Thomas E, Subramanian G, Keiser P, Moore TA. Treatment of patients with refractory giardiasis. Clin Infect Dis. 2001 Jul 1;33(1):22-8. doi: 10.1086/320886. Epub 2001 May 23. PMID 11389490
- [Derived] Corda M, Sciurba J, Blaha J, Mahanty S, Paredes A, Garcia HH, Nash TE, Nutman TB, O'Connell EM. A recombinant monoclonal-based Taenia antigen assay that reflects disease activity in extra-parenchymal neurocysticercosis. PLoS Negl Trop Dis. 2022 May 26;16(5):e0010442. doi: 10.1371/journal.pntd.0010442. eCollection 2022 May. PMID 35617367
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1997-I-0096.html